CLINICAL TRIAL: NCT04112017
Title: A Multicenter, Randomized, No-treatment Controlled, Parallel, Evaluator-blind, Medical Device Pivotal Study to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 360 Injected Into Dorsal Hand for Hand Augmentation to Correct Volume Loss
Brief Title: A Study of YVOIRE Y-Solution 360 for Hand Augmentation to Correct Volume Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL019
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Dorsal Hand Volume Loss
Keywords: Hyalunic acid; Filler; Dorsal hand; Medical device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YVOIRE Y-Solution 360 (Experimental): Maximum 5 ml including touch-up
  Interventions: Device: YVOIRE Y-Solution 360
- No-treatment (No Intervention): No-treatment. At 12 weeks after the assessment, treatment maximum 5 ml including touch-up

INTERVENTIONS:
Device: YVOIRE Y-Solution 360 — Hyaluronic acid
  Arms: YVOIRE Y-Solution 360

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of YVOIRE Y-Solution 360 in the treatment of dorsal hand to correct volume loss.

ELIGIBILITY:
Inclusion Criteria:

1. 19 Years and older
2. Hand Volume Rating Scale (HVRS) of grade 2 or 3 with both hands
3. Participants who are willing to undergo the treatment of dorsal hand to correct volume loss

Exclusion Criteria:

1. Congenital defect, external injuries, lipodystrophy, unhealed wound, disease related-abnormalities, or tumors on the dorsal hands
2. Active inflammation or infection on the dorsal hands
3. Received anti-coagulation therapy, anti-platelet therapy, or expected to require repeated treatment within 2 weeks prior to visit 2 (randomization)
4. Had locally applied ointments (steroid, retinoid, anti-wrinkle production, tanning, or any other form of irritating product) or expected to require repeated treatment within 4 weeks prior to visit 2 (randomization)
5. Received immuno-suppressive medication including systemic glucocorticoids or expected to require repeated treatment within 8 weeks prior to visit 2 (randomization)
6. Received NSAIDs, Vitamin E, or expected to require repeated treatment within 1 week prior to visit 2 (randomization)
7. Had dermal filler injections (HA, CaHA, silicon, PAAG, PMMA etc.), Botulinum toxin therapy, adipose tissue transplantation, or esthetic surgery within 12 months prior to visit 2 (randomization)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
≥ 1 grade improvement on Hand Volume Rating Scale (HVRS) as assessed by the evaluator-blinded | 12 weeks after treatment
  5-grade photonumeric hand grading scale (grade 0 - grade 4)

SECONDARY OUTCOMES:
≥ 1 grade improvement on Hand Volume Rating Scale (HVRS) as assessed by the evaluator-blinded and the treating investigator | Up to 52 weeks after treatment
  5-grade photonumeric hand grading scale (grade 0 - grade 4)
≥ 1 grade improvement on Global Aesthetic Improvement Scale (GAIS) as assessed by the treating investigator and the subject | Up to 52 weeks after treatment
  5-point scale rating global aesthetic improvement in appearance (score -1 - score 3)
Change from baseline on Hand Volume Rating Scale (HVRS) as assessed by the evaluator-blinded and the treating investigator | Up to 52 weeks after treatment
  5-grade photonumeric hand grading scale (grade 0 - grade 4)
Change from baseline on Global Aesthetic Improvement Scale (GAIS) as assessed by the treating investigator and the subject | Up to 52 weeks after treatment
  5-point scale rating global aesthetic improvement in appearance (score -1 - score 3)
Safety profile as assessed by incidence of adverse events | Up to 52 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Soonchunhyang University, Bucheon-si, Gyeonggi-do
  - Eulji Hospital, Seoul